CLINICAL TRIAL: NCT05454228
Title: Relationship Between Neuroinflammatory Biomarkers and Postoperative Delirium in Elderly Patients With Hip Replacement
Brief Title: Biomarkers and Postoperative Delirium in Elderly Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: biomarkers
Record Dates: First submitted 2022-06-07; First posted 2022-07-12 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-06

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delirium
  Interventions: Behavioral: postoperative delirium
- Non-delirium
  Interventions: Behavioral: postoperative delirium

INTERVENTIONS:
Behavioral: postoperative delirium — Postoperative delirium (POD) occurs within 1 week after surgery in patients, with obvious time characteristics, mainly occurring within 1-3 days after surgery. Postoperative delirium has adverse effects on the short and long term prognosis of patients. Patients with delirium have an increased risk of postoperative complications, perioperative death, longer hospital stay and increased medical costs during hospitalization.

SUMMARY:
This study intends to verify and explore the correlation of neuroinflammation biomarkers in cerebrospinal fluid and plasma of elderly patients undergoing hip replacement with postoperative delirium, so as to achieve a new method to predict whether patients will develop postoperative delirium and improve the prognosis of elderly patients with postoperative delirium. Reduce the probability of postoperative complications, improve the long-term survival rate of patients after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. age≥65
2. Patients undergoing hip replacement under spinal anesthesia
3. ASA grade I~III;
4. Voluntarily participate in this study, and informed consent was signed by the patients themselves and their families

Exclusion Criteria:

1. Patients with multiple fractures and trauma
2. Patients with preoperative cognitive dysfunction determined by MMSE scale;
3. Severe impairment of hearing, visual and language system functions;
4. Not suitable for or unwilling to undergo subarachnoid anesthesia
5. Patients who refuse to participate or cannot cooperate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients undergoing hip replacement surgery in Henan Provincial People's Hospital were selected during the trial
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
neuroinflammatory biomarkers | preoperative、24 hours after surgery、48 hours after surgery
  Whether there are changes in neuroinflammatory biomarkers(Ykl40(pg/mL), procalcitonin(ng/mL), IL-17A,IL-23,INF-γ(IU), Tau(pg/mL), amyloid beta(pg/mL),etc) in cerebrospinal fluid and plasma between delirium patients and non-delirium patients before and after operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan People's Hospital, Zhengzhou, Henan, China